CLINICAL TRIAL: NCT03867175
Title: A Randomized Trial of Consolidative Immunotherapy With vs Without Thoracic Radiotherapy and / or Stereotactic Body Radiation Therapy (SBRT) After First-Line Systemic Therapy for Metastatic NSCLC
Brief Title: Immunotherapy With or Without SBRT in Patients With Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056681; NCI-2019-01259 (Other: Clinical Trial Reporting Program); CCCWFU 62718 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Lung Cancer; Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab (Experimental): 3-10 treatments of SBRT/ pembrolizumab IV for 30 minutes every 3-4 weeks for 1 year at doctor's discretion.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Biological: Pembrolizumab
- Arm 2 Pembrolizumab Only (Experimental): Patients receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Patients undergo 3-10 treatments of stereotactic body radiation therapy (SBRT)
  Other Names: Stereotactic Ablative Body Radiation Therapy
  Arms: Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab
Biological: Pembrolizumab — Patients undergo 3-10 treatments of SBRT. Patients also receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase III trial studies immunotherapy and stereotactic body radiation therapy to see how well it works compared with immunotherapy alone after first-line systemic therapy (therapy that goes throughout the body) in treating patients with stage IV non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving immunotherapy with stereotactic body radiation therapy may work better than immunotherapy alone in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival of patients randomized to radiation and consolidative immunotherapy against those receiving consolidative immunotherapy alone.

SECONDARY OBJECTIVES:

I. To estimate overall survival in all patients and will compare overall survival of those randomized to radiation and consolidative immunotherapy against those receiving consolidative immunotherapy alone.

II. In patients receiving radiation, to describe the rate of in-field local control and rate of out-of-field disease progression with serial imaging.

III. In patients not receiving radiation, describe progression at known sites of disease after first line systemic therapy and rate of development of new metastases with serial imaging.

IV. To evaluate toxicity associated with radiation followed by consolidative immunotherapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo 3-10 treatments of stereotactic body radiation therapy (SBRT). Patients also receive pembrolizumab intravenously (IV) over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.

ARM II: Patients receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 1 year, every 6 months for the next 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older.
* Performance Status 0-2 (ECOG) at time of consult with radiation oncology.
* Pathologically proven non-small cell lung cancer (NSCLC) with evidence of metastatic disease.
* Must have received 4 cycles of standard of care systemic therapy (usually this will consist of combination chemo-immunotherapy), with a CT chest abdomen pelvis that was performed after completion of these 4 cycles and demonstrates no evidence of progression per RECIST v1.1.
* To be eligible for enrollment and randomization, patients must be within 180 days from their first dose of standard of care systemic therapy. Cycle 1 day 1 is defined as day 1. If enrolled on day 180, the patient would need to be randomized the same day.
* Persistent active disease must be amenable to radiation treatment per the treating radiation oncologist, and patients must have at least one residual site of disease which can be identified by CT or PET/CT and targeted with radiation.
* Patients who previously had earlier stage NSCLC treated definitively and have now developed new distant disease, are eligible for inclusion if they have undergone at least 4 cycles of standard of care systemic therapy for their metastatic recurrence, and they meet all criteria above.
* There are no strict size or tumor number limitations in a given organ (lung, liver, abdomen pelvis, or spine). This is at the discretion of the treating radiation oncologist.

Exclusion Criteria from Enrollment

* More than 180 days has elapsed since day 1 of cycle 1 of standard of care systemic therapy.
* Pregnant or lactating women.
* The patient has received treatment for other carcinomas within the last three years (Except for cured non-melanoma skin cancer, low-risk prostate cancer, T1/T2 glottic cancer, stage 0 or stage I breast cancer, non-invasive bladder cancer, or treated in-situ cervical cancer). Prior lung cancer diagnosis now with oligometastatic recurrence is not an exclusion criteria.
* Patients with major activating mutations in EGFR (del19, L858R, and T790M) or ROS 1 or ALK gene rearrangements are excluded

Eligibility for Randomization

* Once enrolled on study, patients will have a PET/MRI brain for restaging. Patients with no evidence of progression and 8 or fewer sites of active persistent disease per the treating physician are eligible for randomization.
* If a PET has been performed within 30 days of enrollment with no evidence of progression per RECIST v1.1, then this scan may be used and does not have to be repeated prior to randomization.
* If an MRI brain has been performed within 90 days of enrollment with no evidence of progression per RECIST v1.1, then this scan may be used and does not have to be repeated prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.9) | 53 | 59.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (PFS) After Completion of First Line Standard of Care Systemic Therapy
Description: Will be determined using the product-limit method of Kaplan and Meier. Will compare unadjusted median PFS between the 2 arms using a log-rank test. Will also use a proportional hazards model to compare progression-free survival between the two groups, adjusting for key covariates such as age, performance (Eastern Cooperative Oncology Group) status, response to initial systemic therapy versus (vs) stable disease, the presence or absence of brain metastases, PD-L1 [programmed death-ligand ] expression (< 1% vs > 50%), tumor histology (adenocarcinoma vs non-adenocarcinoma), and number of disease sites treated (1-3 sites vs 4-6 sites). Progression is defined using RECIST v1.1 is relative Increase: A 20% increase in the sum of the longest diameters of target lesions (from baseline or nadir) is a criterion for PD.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab: 3-10 treatments of SBRT/ pembrolizumab IV for 30 minutes every 3-4 weeks for 1 year at doctor's discretion.
  There were 4 participants in Arm 1. One person progressed (date of progression, 1/8/2020; date of death 2/18/2020; study start date 6/24/2019).
  The remaining 3 are censored (no progression, no death) and still alive as of April 23, 2025.
- Arm 2 Pembrolizumab Only: Patients receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.
  The one participant in this arm is alive and censored (no progression, no death) as of April 23, 2025.
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

2. Secondary Outcome: Number of Participants With Overall Survival
Description: Overall Survival is defined as the duration from the start of first line standard of care systemic therapy to the date of death or date of last contact; those lost to follow-up will be censored and will be reported with an exact 95% confidence interval.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab: 3-10 treatments of SBRT/ pembrolizumab IV for 30 minutes every 3-4 weeks for 1 year at doctor's discretion.
  There were 4 participants in Arm 1. One person died (date of death 2/18/2020; study start date 6/24/2019). The remaining 3 are censored (no progression, no death) and still alive as of April 23, 2025.
- Arm 2 Pembrolizumab Only: Patients receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.
  The one participant in this group is alive and censored (no progression, no death) as of April 23, 2025.
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Progression
Description: In patients not receiving radiation, the investigators will assess progression at their known sites of disease prior to beginning first line systemic chemotherapy.
Time Frame: Baseline up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

4. Secondary Outcome: Number of Participants to Have a Rate of Failure
Description: Investigators will assess the rate of failures inside and outside of radiation treatment.
Time Frame: Baseline up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

5. Secondary Outcome: Number of Participants With New Sites of Disease
Description: Investigators will assess the development of new sites of disease during or after immunotherapy
Time Frame: Baseline up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab: 3-10 treatments of SBRT/ pembrolizumab IV for 30 minutes every 3-4 weeks for 1 year at doctor's discretion.
  The one patient in Arm 1 who had progression had progression in a new site of disease.
  No other patients in Arm 1 had progression.
- Arm 2 Pembrolizumab Only: Patients receive pembrolizumab IV over 30 minutes every 3-4 weeks for 1 year at the discretion of the treating physician.
  The one patient in Arm 2 had no progression.
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Adverse Events
Description: All safety measures, including acute and late toxicity, will be reported using descriptive statistics (mean, median, standard deviation, proportions, and 95% confidence intervals). This will include calculating frequency/risk of adverse events by treatment site. Potential toxicities reported would include pneumonitis, esophagitis, chest wall pain, dermatologic toxicity, renal dysfunction, gastrointestinal toxicity including nausea, vomiting, and diarrhea, hepatotoxicity, and abdominal pain. These toxicities would be assessed according to site of irradiation by the treating physician and graded as per Common Terminology Criteria for Adverse Events 5.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
Number analyzed (Participants) | 4 | 1
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab | Arm 2 Pembrolizumab Only
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab (N=4) | Arm 2 Pembrolizumab Only (N=1)
Hypertension (Vascular disorders) | 2 (6) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Stereotactic Body Radiation Therapy/Pembrolizumab (N=4) | Arm 2 Pembrolizumab Only (N=1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (6) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (6) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study enrolled n=5 patients. Four of 5 were randomized to arm 1, and the remaining patient was randomized to arm 2.

Only one patient (arm 1) had any primary/secondary outcomes--1 patient in arm 1 had progression to a new disease site and died soon thereafter.

Due to these small numbers statistical analysis (e.g., rates, statistical comparisons of arms) are not possible.

Descriptive and count data have thus been entered into the outcomes data fields.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03867175/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT03867175/ICF_001.pdf